CLINICAL TRIAL: NCT00133666
Title: Improving Asthma Communication in Minority Families
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Arlene Butz, ScD, RN, Johns Hopkins University, Department of Pediatrics
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 03-11-11-05
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2008-07-17 (Estimated); Status verified 2008-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Asthma Communication Education
- 2 (Active Comparator)
  Interventions: Behavioral: Standard Asthma Education

INTERVENTIONS:
Behavioral: Asthma Communication Education
  Arms: 1
Behavioral: Standard Asthma Education
  Arms: 2

SUMMARY:
The purpose of this study is to determine if teaching children with asthma how to talk to their doctor about controlling their asthma including symptom frequency in an asthma diary and medication use techniques, will result in less symptom and missed school days, fewer emergency room visits and reduce the cost of asthma health care.

DETAILED DESCRIPTION:
Children with persistent asthma are often not receiving regular preventive asthma care despite experiencing frequent asthma symptoms. When linked to timely and appropriate asthma medication use, good physician-parent-child communication is associated with a decrease in asthma morbidity and mortality. Removing obstacles to preventive asthma care and improving communication between the parent-children and PCP are two necessary prerequisites to improving asthma outcomes in low-income minority children.

We, the researchers at Johns Hopkins University, hypothesize that a culturally-tailored parent and child asthma communication intervention (ACI) designed to teach parent and child communication skills for use with their health care provider regarding asthma symptom severity, medication use, personal goal of treatment and quality of life issues will significantly reduce emergency room utilization for asthma care. We propose to compare this parent/child asthma communication intervention (ACI) to a developed standard asthma education intervention (SAE) designed to increase basic asthma self-management.

This study will advance nursing science by improving asthma self-management for school age children, who may be self-administering their asthma medications, yet not participate in receiving information or making their own medical decisions regarding their asthma. The proposed study is targeted at low-income minority school-aged children with evidence of poorly controlled, high-risk asthma. If successful, this intervention could have significant practical applications as a component of asthma nurse-case management, to practice currently being employed by many managed care groups across the country as an intervention for their high-risk/high ED use asthma patients. Because of the high prevalence and enormous health impact of asthma and the disproportionate asthma burden experienced by minority children, the outcome of the proposed study will have significant pediatric nursing applicability.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-12 years
* Physician diagnosis of asthma
* Reside in metropolitan Baltimore
* English speaking
* Able to read 80% of parent educational brochure in English
* Emergency Department (ED) visit within the past 12 months and can identify a primary care provider
* No other co-morbid pulmonary disease

Exclusion Criteria:

* Enrolled in another asthma study

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 231 (Actual)
Dates: Start 2004-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Reduce the cost of asthma health care. | 18 Months

SECONDARY OUTCOMES:
Fewer emergency room visits | 18 Months
Less symptoms | 18 Months
Fewer missed school days | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Butz, SCD,MSN,BSN, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Logan J and Butz AM. Improving asthma communication in minority families - ongoing pilot study. Am J Respir and Crit Care Med. 2004; Abstract No. 5119, American Thoracic Society International Meeting, Orlando, FL, May 2004. Butz AM. Effective asthma communication: Children and primary care providers. European Respiratory Society Annual Congress. September 2004, Glasgow, Scotland.
- [Derived] Butz A, Kub J, Donithan M, James NT, Thompson RE, Bellin M, Tsoukleris M, Bollinger ME. Influence of caregiver and provider communication on symptom days and medication use for inner-city children with asthma. J Asthma. 2010 May;47(4):478-85. doi: 10.3109/02770901003692793. PMID 20528605